CLINICAL TRIAL: NCT04229277
Title: Fast Track Diagnosis of Skin Tumours by Four Different Advanced Imaging Technologies - a Clinical Study
Brief Title: Fast Track Diagnosis of Skin Cancer by Advanced Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Mette Mogensen, MD, PhD, Ass. Prof., Chief Consultant, University Hospital Bispebjerg and Frederiksberg
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: H-19036900
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Malignant Melanoma; Nevus, Pigmented; Basal Cell Carcinoma; Seborrheic Keratosis
MeSH Terms: conditions — Melanoma; Nevus, Pigmented; Carcinoma, Basal Cell; Keratosis, Seborrheic | interventions — Tomography, Optical Coherence; Ultrasonography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- in tumours (Other): consecutive enrollment of newly referred skin tumour patients
  Interventions: Diagnostic Test: optical coherence tomography

INTERVENTIONS:
Diagnostic Test: optical coherence tomography — comparison of four imaging technologies in skin tumour diagnosis
  Other Names: photoacoustic imaging; in vivo confocal microscopy; doppler ultrasound

SUMMARY:
Aim of study:

To collect data for a new image-guided diagnostic algoritm, enabling the investigators to differentiate more precisely between benign and malignant pigmented tumours at the bedside. This study will include 60 patients with four different pigmented tumours: seborrheic keratosis (n=15), dermal nevi (n=15), pigmented basal cell carcinomas (n=15), and malignant melanomas (n=15), these four types of tumours are depicted in Fig.1, and all lesions will be scanned by four imaging technologies, recruiting patients from Sept 2019 to May 2020. In vivo reflectance confocal microscopy (CM) will be used to diagnose pigmented tumours at a cellular level and provide micromorphological information5;6. Flourescent CM will be applied to enhance contrast in surrounding tissue/tumours. Optical coherence tomography (OCT), doppler high-frequency ultrasound (HIFU) and photoacustic imaging (also termed MSOT, multispectral optoacustic tomography) will be used to measure tumour thickness, to delineate tumours and analyze blood flow in blood vessels. Potential diagnostic features from each lesion type will be tested. Diagnostic accuracy will be statistically evaluated by comparison to gold standard histopathology

DETAILED DESCRIPTION:
Study design The prospective non-blinded clinical study will include with seborrheic keratosis (n=15), dermal nevi (n=15), pigmented or dark basal cell carcinomas (n=15), and malignant melanomas (n=15) referred to or diagnosed at Dept. of Dermatology, Bispebjerg Hospital. All tumours are histologically verified by skin biopsy. To explore clinical feasibility and diagnostic accuracy of four different skin imaging technologies all patients will be scanned by an experienced examiner in one 2-hour session. If patients demonstrate more than one skin tumour within the same anatomical location, all lesions will be included and scanned. Lesions in other anatomical areas of the same patient will not be included. The total extra time spend in the department to participate in this study will be approximately 2-3 hours for each patient. Only one visit is required to participate. The skin tumors in patients enrolled will subsequently be treated according to hospital and national guidelines.

Background: A bedside examination of a skin tumours using advanced imaging technology is considered a valuable future tool for Dermatologists. The investigators vision is to provide image guided skin cancer therapy to all patients with skin tumours. This study compares clinical feasibility and diagnostic accuracy of four different imaging technologies applied in a fast-track bedside analysis of various skin tumours; four different types, 2 benign and 2 malignant types.

It is also hypothesized that:

* Due to higher resolution UHR-OCT may have higher diagnostic accuracy than C-OCT.
* Doppler HIFU and optoacustic imaging diagnosis may be more accurate in skin tumours thicker than 1-2 mm compared to diagnosis based on OCT imaging.
* The cellular resolution of RCM and the detailed blood flow information acquired from photoacustic imaging may supplement clinical decision making and increase diagnostic accuracy compared to only OCT or only HIFU.

Study objectives

Primary objective:

This study explores the clinical utility of four skin imaging technologies: scanning time, clinical feasibility (does the skin tumour fit into the scanning probe) and diagnostic accuracy. The investigators examine patients with four different common skin tumour types referred to Dept of Dermatology, BFH using four different advanced imaging technologies; five different tools as investigators apply two different OCT-systems.

Secondary outcome measures:

* To measure diagnostic accuracy of index tests (OCT, RCM, HIFU and photoacoustic imaging)
* To measure tumor size by OCT, photoacoustic imaging and HIFU
* To explore if UHR-OCT detects features in tumors that C-OCT cannot detect.
* To explore if information from dynamic C-OCT images of dermal blood vessels inside the skin tumour increases diagnostic accuracy
* To explore if information from doppler ultrasound images of dermal vessels inside the tumour increases diagnostic accuracy
* To explore if information from photoacoustic imaging of dermal vessels inside the tumour increases diagnostic accuracy
* To report potential decreased time delay from first visit to efficient skin cancer treatment
* To record survival rates
* To record treatment types and number of therapeutic sessions (e.g. operations)
* To report potential adverse device events
* To report patient satisfaction of scanning procedures

Evaluation of skin tumours All skin tumours will be evaluated clinically, by two different OCT systems (C-OCT and UHR-OCT), by RCM, by photoacoustic imaging and doppler HIFU. Skin biopsies will be performed according to standard hospital procedures. Skin punch biopsies from skin tumours are required for treatment planning and is not part of this research project. Accordingly, a skin biopsy will be performed as part of the treatment plan independent of whether the patient is recruited or not.

Imaging Technologies In vivo reflectance confocal microscopy (CM) will be used to diagnose pigmented tumours at a cellular level and provide micromorphological information5;6. Flourescent CM will be applied to enhance contrast in surrounding tissue/tumours. Optical coherence tomography (OCT), doppler high-frequency ultrasound (HIFU) and photoacustic imaging (also termed MSOT, multispectral optoacustic tomography) will be used to measure tumour thickness, to delineate tumours and analyze blood flow in blood vessels. Potential diagnostic features from lesion types will be tested. Diagnostic accuracy will be statistically evaluated by comparison to gold standard histopathology The imaging methods OCT, RCM and doppler ultrasound, are technologies that are routinely used in the clinic at Dept of Dermatology, BFH and all investigators are highly trained in using the scanners. The UHR-OCT is a prototype and the photoacoustic system is a brand-new clinical device. OCT, RCM and ultrasound examinations are performed in a darkened room. The images of all patients will be saved in a digital archiving computer system for subsequent scoring and further evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. 60 Patients with histologically verified: seborrheic keratosis 15 in total, dermal nevi 15 in total, pigmented BCC in total, and malignant melanomas 15 in total on areas of the body where scanning is feasible with all five systems
2. Patients with skin tumours clinically suspicious of one of the four lesions mentioned in (1), that are not yet biopsied, if the patient is willing to undergo a skin biopsy from the suspicious lesion
3. > 18 years of age at baseline
4. Legally competent, able to give verbal and written consent
5. Communicate in Danish verbally as well as in writing
6. Subject in good general health, is willing to participate and able to give informed consent and can comply with protocol requirements.

Exclusion Criteria:

1. Individuals with other skin diseases in the skin area of interest
2. Individuals who´s skin tumour is not accessible for imaging e.g. inside the ear, inside nostrils, on eyelids
3. Subjects who will not undergo a skin biopsy after imaging of the suspicious tumour clinically diagnosed as BCC
4. Pregnancy
5. Women of child-bearing potential not using a contraceptive agent at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of the four methods imaging methods compared to histopathology of skin tumours. | 6-12 months
  Sensitivity is expressed in percentage and defines the proportion of true positive subjects with the disease in a total group of subjects with the disease (TP/TP+FN). Sensitivity is defined as the probability of getting a positive test result in subjects with the disease (T+|B+). Specificity is a measure of diagnostic test´s accuracy, complementary to sensitivity. It is defined as a proportion of subjects without the disease with negative test result in total of subjects without disease (TN/TN+FP). Sensitivity and specificity are reported in percent

SECONDARY OUTCOMES:
tumour thickness | 6-12 months
  in millimeters
survival rates | 12 months
  in number of months
blood flow in skin tumours | 6-12 months
  expressed in arbitrary units in OCT volume scans and in volume densities/second in doppler ultrasound images
To report potential decreased time delay from first visit to efficient skin cancer treatment | 12 months
  Expressed as duration of time from diagnosis till initial treatment in number of days
To record treatment types and number of therapeutic sessions (e.g. operations) | 12 months
  For each study participant treatment types are listed in numerical numbers and so is the number of treatment sessions counted and listed for each individual participant in this trial
To report patient satisfaction of scanning procedures | 6-12 months
  A questionnaire with qualitative questions (How did you like being scanned?) and quantitative questions: on a scale from 0-10 how painful was the scanning procedure)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Dermatology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The images file data will be very large and will be situated on the hospital server. We cannot legally share these files.